







Research Protocol: Online guided self-help intervention for sexual distress following sexual assault: A single case experimental study

#### **PROTOCOL**

# <u>Title:</u> Online guided self-help intervention for sexual distress following sexual assault: A single case experimental study

Short Title: Guided Self Help Following Sexual Assault: SCED

IRAS Project ID: 313482

#### **Sponsor:**

Royal Holloway, University of London Egham, Surrey TW20 0EX

#### **Chief Investigator:**

Kimberley Khoo Doctorate in Clinical Psychology, Department of Psychology Royal Holloway, University of London Egham, Surrey TW20 0EX

Telephone: +44 07492418618 Email: njjt001@live.rhul.ac.uk

## **Supervisors:**

Andy Macleod

Director

Doctorate in Clinical Psychology

Royal Holloway, University of London

Egham, Surrey

**TW20 0EX** 

Email: A.Macleod@rhul.ac.uk

Jane Vosper

Clinical Psychologist

Doctor of Clinical Psychology (DClinPsy)

Barts Health NHS Foundation Trust

Sexual Wellbeing Service

Grahame Hayton Unit Ambrose King Centre Royal London Hospital,

Whitechapel

E1 2BB

Email: jane.vosper3@nhs.net

V2 10/10/22

2

# Contents

| Sy | nopsis study | 5 |
|----|---------------------------------------------------|----|
| • | 1. Background and rationale | |
| | 1.1 Need for research in this area | |
| | 1.2 Aims | 6 |
| | 1.3 Objectives. | 7 |
| | 2. Methods | 7 |
| | 2.1 Study design. | 7 |
| | 2.2 Recruitment and participant screening | 8 |
| | 2.2.1 Inclusion criteria | 11 |
| | 2.2.2 Exclusion criteria | 11 |
| | 2.2.3 Criteria for premature withdrawal | 12 |
| | 2.3 Materials provided to participants | 12 |
| | 2.3.1 Intervention | 12 |
| | 2.3.2 Visual Analogue Scales | |
| | 2.3.3 Female Sexual Dysfunction Scale | 13 |
| | 2.3.4 Female Sexual Functioning Index | 14 |
| | 2.3.5 State Self Compassion Scale | 14 |
| | 2.3.6 Client Satisfaction Questionnaire | 14 |
| | 2.3.7 Feedback form | 14 |
| | 2.4 Expert by experience involvement | 15 |
| | 3. Study procedure | |
| | 3.1 Informed consent procedures | 16 |
| | 3.2 Data collection methods | 16 |
| | 3.3 Statistical analysis of data | 17 |
| | 3.4 Risk and burdens | |
| | 3.5 Study end definition | 19 |
| | 3.6 Pause criteria for study | |
| | 4. Assessment of safety | |
| | 5. Data security management and confidentiality | |
| | 5.1 Data storage and handling and confidentiality | 20 |
| | 5.2 Data preservation | 21 |
| | 6 Publication of results | 21 |

# **Study Synopsis**

| Full Title | Online guided self-help intervention for sexual distress following sexual assault: A single case experimental study |
|---|---|
| Short Title | Guided self-help following sexual assault - SCED |
| Protocol version number and date | V2 250722 |
| Study duration | 10 months |
| Study design | Single Case Experimental Design |
| Sponsor | Royal Holloway, University of London |
| Chief Investigator | Kimberley Khoo |
| IRAS Project ID | 313482 |
| Primary objective | To test the acceptability and feasibility of an online guided self-help intervention by female survivors of sexual assault who experience sexual distress |
| Secondary objective | To gain an initial indicator on the effectiveness of the intervention |
| Number of subject | 6 |
| Main inclusion criteria | Cis-female over the age of 18 with an experience of sexual assault that occurred over 12 months ago |
| Statistical methodology and analysis | Descriptive statistics, visual analysis, reliable change index. |

1. Background & Aims of the project

1.1 Need for research in this area

Sexual assault (SA) is associated with enduring negative impacts, including interpersonal,

psychological and physical difficulties (Maniglio, 2009; Chen et al., 2010). SA survivors

develop a different relationship with sex (O'Callaghan et al., 2018) and report less interest in

sex, reduced desire, fear of sex, arousal dysfunction and painful sex (Norris & Feldman-

Summers, 1981; Weaver, 2009). They also experience high levels of shame, self-blame and

decreased self-compassion and attachment-based difficulties (Hamrick & Owen, 2019).

Despite the prevalence of these difficulties, there is limited research identifying treatment.

Systematic reviews investigating the effectiveness of psychological interventions in SA

survivors do not mention sexual distress, suggesting that interventions are limited or do not

consider sexual distress (Regehr et al., 2013; Parcesepe et al., 2015). Instead, they target

generic distress related to trauma. Evidence from a meta-analysis suggests that psychological

treatments for post-traumatic stress disorder following SA had no effect on sexual problems

(O'Driscoll & Flanagan, 2015). On the other hand, traditional psychosexual therapy that aim

to alleviate sexual distress does not consider the experience of SA trauma symptoms and how

they may interact with standard psychosexual approaches (Althof et al., 2005). Meston and

colleagues (2013) found that standard psychosexual therapy developed to alleviate sexual

difficulties had inconsistent results among women with a history of SA, suggesting precedence

for developing specific psychosexual intervention for SA survivors. Few studies explored

specific interventions for sexual distress experienced by SA survivors; however, most of these

studies do not adopt a formal model or follow a standard protocol (Gerwitz-Meydan, 2020).

V2 10/10/22 IRAS: 313482

This study proposes an online four-session guided self-help psychoeducational program for

survivors of SA. Online guided-self-help is the chosen modality as it widens access to treatment

in a population who may experience shame and stigma regarding help-seeking (Levin et al.,

2018). Previous studies, such as a pilot RCT found online guided self-help effective in

improving sexual functioning in women with vaginismus (Zarski et al., 2017). A treatment

protocol for Internet-based guided self-help has already been developed for sexual pain but not

for sexual distress after SA (Zarski et al., 2018). This intervention aims to normalise and build

women's confidence on getting back to sex after experiencing SA. The objective is to reduce

shame, self-criticism, sexual distress and improve sexual well-being. By exploring an

individual's difficulties through a normalising framework, the intervention aims to increase

their awareness of their difficulties and build confidence, skill and motivation to alleviate

sexual distress. As this is a novel intervention, the study adopts a single-case experimental

design (Morley, 2017). It aims to test the acceptability and feasibility and potential

effectiveness of the intervention.

To our knowledge, no research projects have developed guided self-help materials for female

survivors of sexual abuse targeting sexual distress. The project has taken guidance from experts

by experience to develop materials collaboratively. Clinical psychologists from Bart's NHS

Trust Sexual Wellbeing Service, where similar materials have been used in a group setting

have also provided feedback.

**1.2 Aims** 

- To investigate the feasibility and acceptability of a 4-session guided self-help

psychosexual intervention for survivors of sexual abuse

- Initial indicator of effectiveness in reducing sexual distress

V2 10/10/22 IRAS: 313482

2 10/10/22

- Improving sexual satisfaction- specifically confidence in practicing strategies that will

improve their relationship and experience of sex

1.3 Study objectives

Primary objectives

a. The objective of the study is to investigate the feasibility and acceptability of a 4-

session guided self-help intervention for female survivors of sexual assault to gather an

initial indicator of effectiveness in reducing sexual distress.

b. Is the intervention viewed as acceptable by female survivors of sexual assault? We will

be defining 'acceptability' as how willing participants are to use the materials and its

content (Bowen et al., 2009).

Secondary objectives

The secondary outcomes are whether the study suggest the intervention is effective. Is there

an initial indicator that the intervention effective? Effectiveness is measured by reduction in

the measure of sexual distress and improvement of sexual satisfaction – specifically confidence

and motivation in practicing strategies that will improve their experience of sex.

2. Methods

2.1 Study design

The study adopts a single-case experimental design (SCED). This study design is helpful in

testing the novelty and feasibility of an intervention.

Potential participants will be invited to follow a link to a Qualtrics survey. The Qualtrics survey

provides detailed information about the study. Participants will undergo screening for

eligibility and risk via Qualtrics. Should individuals wish to participate and are eligible, they

can give informed consent by reading a set of statements on Qualtrics relating to the study

IRAS: 313482

V2 10/10/22 7

information. Eligible participants will fill in questionnaires such as the FSDI, FSFI, SCSS-S,

at this point. Participants will undergo a baseline period known as phase A, varying between

5- 14 days where they will fill in visual analogue scales daily. The number of days participants

will be in baseline will be randomly allocated by a randomiser. There are 6 visual analogue

scales measuring shame, guilt, self-criticism, self-compassion, normalising and motivation.

After phase A, participants will undergo phase B, which is a 4-week intervention period where

participants go through 1 module of the guided-self-help materials each week and complete the

same visual analogue scales from baseline every day. After phase B, participants will be invited

for a follow-up appointment one month after the intervention to fill in the FSDS, FSFI, client

satisfaction questionnaire (Larsen et al., 1979) and feedback form developed with experts by

experience.

2.2 Recruitment and participant screening

The study will be advertised through Barts NHS Trust Sexual Wellbeing Service with

information put on leaflets circulated within the clinic. Clinicians may also provide an

information sheet to clients with a weblink the study details and screening questionnaire.

Additional recruitment will be done on My Body Back, an organisation who works with

women with experience of sexual assault, in London and Glasgow. My Body Back will

advertise the study on its website and at its events, providing a web link to the study details

and initial screening questionnaire. The intervention will be offered whilst women are on the

waiting list. They will not lose their place on the waiting list if they take part.

General social media advertising will also be done through different charities and communities

who work with female survivors of sexual assault. Potential participants will be encouraged to

take some time to think about whether or not they would like to participate. Individuals will be

V2 10/10/22

8

informed that participation is on a voluntary basis and consent can be withdrawn at any time. They will also not lose their place on the waiting list for services. Statistical power analyses have been underdeveloped for SCED (Arntz et al., 2013). For a SCED, only 1 participant is required for analysis but, Lanovaz & Rapp (2015) suggest a '3 point guideline' as the minimum requirement for control of study design. Having more than 3 participants will also improve the generalization of findings (Kratochwill et al., 2013). Considering this and to account for attrition, we aim to recruit 20 participants with a minimum sample size of 6 participants.

Should individuals wish to participate they will be invited to follow a link to a Qualtrics survey to initial screening questions to check for eligibility. Prior to completing the screening questionnaire participants will be provided the following text 'Thank you for being interested in this study. The next step is to complete a screening questionnaire. This questionnaire aims to determine if this study would be appropriate for you. The questionnaire does not ask you direct questions about your experience of sexual assault; however, it could potentially elicit difficult emotions. Please keep this in mind if you decide to proceed with the questionnaire as your wellbeing is a priority. There are no consequences if you decide to opt out of participating in this study. At the end of the questionnaire, we have included the chief investigator's email along with signposting information about services you can contact if you require additional support. Thank you for your time.' These questions will confirm if participants are experiencing difficulties with sex, have been sexually assaulted over 12 months ago, if they are currently receiving other forms of psychological intervention and have access to a smart phone or computer to access materials. The Patient Health Questionnaire 2-item (PHQ-2) and Generalised Anxiety Disorder 2-item (GAD-2) are incorporated in the screening questionnaire not to screen for depression and/or anxiety but provide an indication of participant demographic. There will also be a risk screen based on the PHQ-9 "Over the past two weeks, V2 10/10/22

how often have you been bothered by thoughts that you would be better off dead or of hurting yourself in some way?" - Not at all, Several days, More than half of the days, Nearly every day and a question about support from family and friends. Those who rate themselves as experiencing thoughts of death or self-harm and do not indicate that they have social support or psychological support will not be eligible to participate (see section. Those ineligible to participate will be redirected to a debrief page, 'debrief page for Qualtrics', which will include an explanation of why this is the case and signposting to relevant resources. They will also be provided with the chief investigators email or given the option to leave their telephone number for the chief investigator to call them and discuss why they were not appropriate for the study. Eligible participants will provide informed consent by reading statements relating to the study information and writing their initials if they consent to each statement. This includes confirming they have read the information, understanding participation is voluntary and being able to withdraw from the research at any time. Participants are asked to provide their GP details as part of informed consent. Participants will be informed that their GP will not be notified about their involvement in the study or provided any information contributed whilst participating. We will only contact their GP if there are identified risks. These risks include increased self-harm behaviour, increased suicidal risk or significant deterioration of mental health. Under these circumstances, confidentiality may be breached and, the chief investigator may contact the participants GP. As there is little to no professional contact as part of the study design, the chief investigator will only be made aware of increased risk if the participant raises it to the chief investigator by email.

Eligible participants who provide informed consent will have a screening call with the lead investigator, Kimberley Khoo to verify risk, confirm consent and answer any additional questions about the study. As the intervention is online, we hope that having a call at the

beginning will increase engagement through the study. After the screening call, participants

will be asked to fill in a participant demographic sheet and provide their name, age, ethnicity,

email address (for contact), region in the UK they live in, employment status and if they are

currently or have previously accessed psychological therapy and what type of therapy they

received. In addition, participants will complete the Female Sexual Distress scale – Revised

(FSDS-R; Derogatis et al., 2002), Female Sexual Function Index (FSFI; Rosen et al., 2000)

and State Self Compassion Questionnaire (SSCS-S; Neff et al., 2021).

2.2.1 Inclusion criteria

- Cis female experiencing sexual distress with a history of sexual trauma

- Willingness to complete guided self help

- Aged 18 and above

- Ability to read English to provide consent and meaningfully engage with the self-help

materials

- Ability to access online guided self-help material through a computer or phone

- Not currently experiencing severe acute mental health problems

- Not currently suicidal or self-harming

2.2.2 Exclusion criteria

Participants will be excluded if they are experiencing severe acute mental health difficulties,

sexual assault occurring within the last 12 months or currently experiencing more than fleeting

suicidal thoughts or engaging in severe self-harming (individuals who have been sexually

assaulted are likely to experience suicidal thoughts or self-harm behaviours, individuals with

fleeting suicidal thoughts or superficial self-harm with strong protective factors may be

V2 10/10/22 IRAS: 313482

included however, since there is no contact with mental health professionals during the

intervention unless participants reach out for triage, it is difficult to assess risk and participants

have to be excluded if they do not have social support systems of are currently accessing

psychological support).

2.2.3 Criteria for premature withdrawal

Participants will be able to withdraw from the study at any point by informing the chief

investigator

2.3 Material provided to participants.

2.3.1 *Intervention* 

4 Sessions of guided self-help will be shared with the participants. These will be in the form of

handout and video recordings that participant access through Qualtrics. The intervention is

based on research on sexual trauma, psychosexual difficulties and materials developed by

Bart's NHS Foundation Trust Sexual Wellbeing Service. It has been made in collaboration

with clinicians within the service, experts by experience and the chief investigator. The

intervention handout and scripts is in the document titled 'Intervention Manual V1'. Within

the document there are scripts for each session which are read out in the video recordings. The

handouts depict the visual images for the video and the materials provided to participant.

Additional handouts for each session can be found in the appendix.

2.3.2 Visual Analogue Scales

Visual analogue scales are to be completed by participants. Visual analogue scales are scales

with two ends where participants will be asked to rate how much they agree or disagree with

the following statements as seen in figure 1 below:

IRAS: 313482

V2 10/10/22 12

#### Shame

o I feel shame when I experience sexual distress

#### Guilt

o I have feelings of guilt when I experience sexual distress

#### • Self-criticism

o When I experience sexual distress, how often do I blame myself or my body?

## Compassion

 When I experience sexual distress, I try to show myself warmth and comfort through my difficulties

#### Normalising

o I understand my difficulties in the context of my experience

#### Motivation

 I am motivated to put things in place to improve/ address the difficulties in my sex life

Figure 1: VAS Example

Disagree

2.3.3 Female Sexual Distress scale – Revised (FSDS-R; Derogatis et al., 2002)

The FSDS-R is used to assess distress related to sex in women (Derogatis et al., 2002). This 13-item self-report questionnaire is scored has four points, (0: never; 1: rarely; 2: occasionally; 3: frequently). In multiple studies involving more than 500 women, the FSDS-R has shown

high internal consistency (Dergostis et al., 2008) for women with and without sexual difficulties. A validation study demonstrate that the measure has discriminant and content validity (Dergostis et al., 2008). The FSDS-R is completed upon recruitment and at the 1 month follow up.

## 2.3.4 Female Sexual Function Index (FSFI; Rosen et al., 2000)

The FSFI is a 19-item questionnaire that measures six domains: desire, arousal, lubrication, orgasm, satisfaction and pain. The questionnaire has been used in different clinical trials and epidemiological studies and have shown to have high test-rested reliability and validity, it is scored from 1 to 5 with different response options. The FSFI is completed upon recruitment and at the 1 month follow up.

#### 2.3.5 State Self Compassion Questionnaire (SSCS-S; Neff et al., 2021)

The SSCS-S is a 6-item questionnaire scored on a 5-point scale from 1 (not very true for me) to 5 (very true for me). In one study, Neff et al (2021) reports the SSCS-S had a strong correlation (r=.96) to the long version of the state self-compassion questionnaire and showed good reliability ( $\alpha = .86$ ). Another study found strong construct validity. The SCSS-S is completed upon recruitment and at the 1 month follow up.

#### 2.3.6 Client Satisfaction Questionnaire (CSQ; Larsen et al., 1979)

The CSQ is an 8-item questionnaire scored on a 4-point scale and will be provided to participants at follow up to ask the acceptability and satisfaction towards the intervention. The questionnaire has high construct validity and internal consistency. Permission has been seeked to adapt the questionnaire to focus on satisfaction for the intervention instead of service satisfaction. Awaiting response. The questionnaire is only used at follow up.

#### 2.3.7 Feedback Form

A short qualitative feedback form will be provided to participants. This form has been developed with experts by experience and will have open ended questions for participants to provide more detailed feedback about the intervention. The questionnaire is only used at follow up.

## 2.4 Expert by experience (EbE) involvement

Survivors of sexual assault were consulted during the development of this study to provide feedback on the session materials and measures used throughout the study. EbE's helped develop the visual analogue scales as well as provide feedback on the intervention scripts and handouts which were implement in the final version.

# 3. Study procedure



Figure 1. Flow chart of study procedures

The study is conducted via Qualtrics, an online survey platform. A survey link will be emailed

to participants for them to complete in their own environment. This allows the study to be

completed anywhere. The survey will be live for 5 months of data collection before being taken

offline. Participants will also be sent handouts of each week's intervention. After completing

the screening questionnaire, eligible participants will be asked to fill in the FSDS-R, FSFI and

SCSS. These questionnaires are filled in once weekly during phase A and B.

During Phase A which varies between 5- 14 days, participants will be sent Qualtrics links to

where fill in visual analogue scales daily. The number of days' participants will be in baseline

will be randomly allocated. There are 6 visual analogue scales that measure shame, guilt, self-

criticism, self-compassion, normalising and motivation.

During phase B participants go through 1 module of the guided-self-help materials each week

and complete the same visual analogue scales from baseline every day. After phase B.

participants will be invited for a follow-up appointment one month after the intervention to fill

in the FSDS, FSFI, SSCS-S client satisfaction questionnaire and feedback form developed with

experts by experience.

3.1 Informed consent procedures

Participants will be asked for informed consent via the Qualtrics survey which states they are

aware of the consequence of taking part in the study and understand the information sheet

provided to them. Participants are also provided with the email address of the Chief

Investigator who they can reach out to with any queries before or after taking part. The study

advertisement will provide brief information about the study. If interested, women will be

directed to the online weblink to read through more detailed study information. It will be clearly

stated that participation is voluntary and participants may drop out at any time and withdraw

consent even after completing the project. It will be clearly stated that the intervention is

Guided Self Help Following Sexual Assault: SCED

provided through online self-help that individuals work through on their own and does not

entail personal support from a psychology team. Through a weblink, participant will tick boxes

to provide informed consent, confirming they consent and understand these terms and asked to

write their name as a way of providing consent.

3.2 Data collection methods

Data collection will be conducted through Qualtrics. During phase A and B, data is collected

daily.

3.3 Statistical analysis of data

Descriptive statistics will be completed for demographic information. Visual analysis will be

performed for daily VAS ratings to evaluate the reliability of treatment effects between the

baseline and treatment phases. To investigate if there is pre-and post-difference between scores

a reliable change index (RCI) will be calculated for each measure using Jacobson & Traux

(1991) to test if changes are statistically significant. Tau-U test will be used on outcomes to

analyse non-overlap of intervention scores. Guidance and procedures will be followed from

What Works Clearing House (Kratochwill et al., 2010).

3.4 Risk and burdens

Participants will not be asked to disclose or directly think about their experience of sexual

assault. The materials developed is to provide psychoeducation and build self-compassion

through a normalising framework that will ask participants to reflect on their sex lives and how

past experiences can affect their experience of sex. This may be difficult and upsetting for some

participants. In order to counter this risk, information and signposting regarding crisis

psychological support will be provided to participants at the beginning and end of each self-

IRAS: 313482

V2 10/10/22

help resource throughout the intervention. Participants will have access to Jane Vosper,

Clinical Psychologist and two other clinicians at the Barts NHS Trust Sexual Wellbeing

Service during the length of project for triage if adverse reactions are identified. Participants

will be able to email the lead investigator and provide consent for the investigator inform Jane

to get in touch with them. Participants will be informed they are able to reach the head

investigator from 9am to 4pm on weekdays. Outside office hours they will be signposted to

other support lines. It will be made clear to participants that besides this one appointment, the

researchers cannot provide further advice or medical treatment

Participants should contact their GPs if they have concerns for their mental or physical health.

Participants are required to provide GP details when providing informed consent. The GP will

not be notified of the participants involvement in the study. We will only contact their GP if

there are identified risk such as severe self-harming, suicidal risk or a significant deterioration

in mental health. Under these circumstances, confidentiality may be breached. As the study is

utilising a self-help intervention, there will be an expectation that participants will be able to

make practical decisions about their readiness to begin the intervention, their ability to cope

and access additional support if required. This expectation will be clearly outlined in the

participant information sheet and consent form.

Participants will be assessed on their risk to self during screening and receive a follow-up

screening call from the head investigator. Participants who disclose high risk who are not

accessing mental health services will be excluded from participating to prevent further distress

that may be triggered during the intervention. Participants will be made aware that the

researcher cannot provide advice or medical treatment and that they should contact their GP as

a first step if they have concerns regarding their mental or physical health. Participants will be

V2 10/10/22 IRAS: 313482

Guided Self Help Following Sexual Assault: SCED

able to provide details of their GP who can be informed that they are taking part in the study,

however this is not compulsory.

Overall, the potential benefits of this study are thought to outweigh the risk. The intervention

content is based on compassion-focused therapy and content that is already used by Barts NHS

trust Sexual Wellbeing Service to improve sexual wellbeing. Participants can access the

materials while waiting to be seen by these services, both of which have a long wait time.

3.5 Study end definition

The study will be considered finished when the statistical analysis has been conducted and

completed as seen as appropriate.

3.6 Pause criteria

If more than 4 participants within eight weeks get in contact with the chief investigator

requesting a 1:1 support session provided by clinicians at Bart's NHS Foundation Trust Sexual

Wellbeing Clinic due to adverse effects from the intervention, the study may be paused. This

number was decided as it represents 25% of our recruitment goal. The study would have to be

paused due to clinician availability. If this occurs, the researchers will have a meeting with the

service lead at Bart's NHS foundation trust Sexual Well-Being Clinic. This meeting will

discuss the feasibility of continuing the study and potentially pausing the study and changing

the recruitment strategy.

4. Assessment of safety

IRAS: 313482

V2 10/10/22 19 As the study is utilising a self-help intervention, there will be an expectation that participants

will be able to make practical decisions about their readiness to begin the intervention, their

ability to cope and access additional support if required. This expectation will be clearly

outlined in the participant information sheet and consent form. Participants will be able to email

the lead investigator and provide consent for the investigator inform Clinicians at Bart's NHS

Foundation trust to get in touch with them. Participants will be informed they are able to reach

the head investigator from 9am to 4pm on weekdays. Outside office hours they will be

signposted to other support lines.

If participants report identified risks, they will be supported through the 1:1 personal support

session provided by Bart's NHS Foundation Trust, Sexual Wellbeing Service. However,

confidentiality may be breached if the clinicians or the chief investigator are still concerned

about risk. The chief investigator will first discuss this with the participant if this occurs.

Subsequently, an urgent email (GP Letter V2) will be sent to the participant's GP via NHS

email. A phone call will also be made to the GP to ensure the GP is informed.

5. Data security, management and confidentiality

5.1 Data storage, handling and confidentiality

All computerised data will be stores and encrypted on a password protected USB drive that

adheres to the NHS confidentiality standards.

Participants will provide email address so that they can be sent links to the self-help materials

each week as well as links to questionnaire and prompt emails. Names are only used when

giving consent and for demographic information. Participants will then be allocated a

participation ID number for reference to fill in questionnaires and not linked to names. A

separate key associating the ID number with the participants' names will be stored apart from

V2 10/10/22 IRAS: 313482

the data and destroyed once it is no longer necessary to contact participants or obtain further

information about them (e.g., once a journal article is published), this file will be password

protected.

All information will be submitted through Qualtrics which is a secure and confidential

platform. Data will be downloaded, password protected and kept on a secure USB stick, only

accessible to the researcher.

Database containing any personal information will be deleted following the final write-up of

the research.

No members of the research team will have access to participants' personal medical records or

any clinical data beyond that voluntarily provided by the participants when they choose to

participate in the study. This information provided will only be seen by the chief investigator

and will be kept securely in a password protected database,

separately to the research data.

Data will be analysed on a personal laptop by the Chief Investigator at Royal Holloway,

University of London. All data will be saved on a password protected encrypted USB

(approved by RHUL and sponsor) that only the chief investigator has access to. This will not

include any personally identifiable data. Data is anonymised and each participant is given a 4-

digit participant code using random numbers and letters.

5.2 Data preservation

The research data will be kept in a database (as discussed in A36) which will be retained by Dr

Andy Macleod, who is supervising this research on behalf of Royal Holloway, University of

London, Data is kept for up to five years, for audit purposes.

This database will contain no personally identifiable information and will be password

protected. Only Dr Andy MacLoed will hold the password. Consent forms will be kept for 2

years.

V2 10/10/22

21

6. Publication of results

The study will be published as a doctoral thesis and may be published in peer reviewed

scientific journals or presented in conferences.

References

Arntz, A., Sofi, D., & van Breukelen, G. (2013). Imagery rescripting as treatment for

complicated PTSD in refugees: a multiple baseline case series study. Behaviour Research and

Therapy, 51(6), 274-283.

Althof, S. E., Leiblum, S. R., Chevret-Measson, M., Hartmann, U., Levine, S. B., McCabe, M.,

... & Wylie, K. (2005). Psychology: Psychological and interpersonal dimensions of sexual

function and dysfunction. The journal of sexual medicine, 2(6), 793-800.

Boersma, K., Håkanson, A., Salomonsson, E., & Johansson, I. (2015). Compassion focused

therapy to counteract shame, self-criticism and isolation. A replicated single case experimental

study for individuals with social anxiety. Journal of Contemporary Psychotherapy, 45(2), 89-

98.

Bowen, D. J., Kreuter, M., Spring, B., Cofta-Woerpel, L., Linnan, L., Weiner, D., ... &

Fernandez, M. (2009). How we design feasibility studies. American journal of preventive

medicine, 36(5), 452-457.

V2 10/10/22

Chen, L. P., Murad, M. H., Paras, M. L., Colbenson, K. M., Sattler, A. L., Goranson, E. N., ...

& Zirakzadeh, A. (2010, July). Sexual abuse and lifetime diagnosis of psychiatric disorders:

systematic review and meta-analysis. In Mayo clinic proceedings (Vol. 85, No. 7, pp. 618-

629). Elsevier.

Derogatis, L. R., Rosen, R., Leiblum, S., Burnett, A., & Heiman, J. (2002). The Female Sexual

Distress Scale (FSDS): Initial validation of a standardized scale for assessment of sexually

related personal distress in women. Journal of Sex & Marital Therapy, 28(4), 317-330.

DeRogatis, L., Clayton, A., Lewis-D'Agostino, D., Wunderlich, G., & Fu, Y. (2008).

Validation of the female sexual distress scale-revised for assessing distress in women with

hypoactive sexual desire disorder. The journal of sexual medicine, 5(2), 357-364.

Gewirtz-Meydan, A. (2020). The relationship between child sexual abuse, self-concept and

psychopathology: The moderating role of social support and perceived parental

quality. Children and youth services review, 113, 104938.

Hamrick, L. A., & Owens, G. P. (2019). Exploring the mediating role of self-blame and coping

in the relationships between self-compassion and distress in females following the sexual

assault. Journal of clinical psychology, 75(4), 766-779.

IRAS: 313482

V2 10/10/22

in oncology, 5, 71.

Jacobson, N. S., & Truax, P. (1991). Clinical significance: A statistical approach to defining meaningful change in psychotherapy research. Journal of Consulting and Clinical Psychology, 59(1), 12 –19.

Jones, S., Ownsworth, T., & Shum, D. H. (2015). Feasibility and utility of telephone-based psychological support for people with brain tumor: a single-case experimental study. Frontiers

Kazdin, A. E. (2019). Single-case experimental designs. Evaluating interventions in research and clinical practice. Behaviour research and therapy, 117, 3-17.

Kratochwill, T. R., Hitchcock, J., Horner, R. H., Levin, J. R., Odom, S. L., Rindskopf, D. M., & Shadish, W. R. (2010). What Works Clearinghouse single-case design technical documentation version 1.0.

Kratochwill, T. R., Hitchcock, J. H., Horner, R. H., Levin, J. R., Odom, S. L., Rindskopf, D. M., & Shadish, W. R. (2013). Single-case intervention research design standards. Remedial and Special Education, 34(1), 26-38.

Larsen, D. L., Attkisson, C. C., Hargreaves, W. A., & Nguyen, T. D. (1979). Assessment of client/patient satisfaction: development of a general scale. Evaluation and program planning, 2(3), 197-207.

Levin, M. E., Krafft, J., & Levin, C. (2018). Does self-help increase rates of help seeking for

student mental health problems by minimizing stigma as a barrier. Journal of American College

Health, 66(4), 302-309.

Manolov, R., Gast, D. L., Perdices, M., & Evans, J. J. (2014). Single-case experimental

designs: Reflections on conduct and analysis. Neuropsychological rehabilitation, 24(3-4), 634-

660.

McLean, L., Steindl, S. R., & Bambling, M. (2018). Compassion-focused therapy as an

intervention for adult survivors of sexual abuse. Journal of child sexual abuse, 27(2), 161-175.

Regehr, C., Alaggia, R., Dennis, J., Pitts, A., & Saini, M. (2013). Interventions to reduce

distress in adult victims of rape and sexual violence: A systematic review. Research on Social

Work Practice, 23(3), 257-265.

Rosen, C. Brown, J. Heiman, S. Leiblum, C. Meston, R. Shabsigh, D. Ferguson, R. D'Agostino,

R. (2000). The Female Sexual Function Index (FSFI): a multidimensional self-report

instrument for the assessment of female sexual function. Journal of sex & marital

therapy, 26(2), 191-208.

Parcesepe, A. M., Martin, S. L., Pollock, M. D., & Garcia-Moreno, C. (2015). The

effectiveness of mental health interventions for adult female survivors of sexual assault: A

systematic review. Aggression and violent behavior, 25, 15-25.

V2 10/10/22

Lanovaz, M. J., & Rapp, J. T. (2016). Using single-case experiments to support evidence-based

decisions: How much is enough?. Behavior Modification, 40(3), 377-395

Maniglio, R. (2009). The impact of child sexual abuse on health: A systematic review of

reviews. Clinical psychology review, 29(7), 647-657.

Meston, C. M., Lorenz, T. A., & Stephenson, K. R. (2013). Effects of expressive writing on

sexual dysfunction, depression, and PTSD in women with a history of childhood sexual abuse:

Results from a randomized clinical trial. The Journal of Sexual Medicine, 10(9), 2177-2189.

Norris, J., & Feldman-Summers, S. (1981). Factors related to the psychological impacts of rape

on the victim. Journal of Abnormal Psychology, 90(6), 562.

Tate, R. L., Perdices, M., McDonald, S., Togher, L., & Rosenkoetter, U. (2014). The design,

conduct and report of single-case research: Resources to improve the quality of the

neurorehabilitation literature. Neuropsychological Rehabilitation, 24(3-4), 315-331.

O'Callaghan, E., Shepp, V., Ullman, S. E., & Kirkner, A. (2019). Navigating sex and sexuality

after sexual assault: A qualitative study of survivors and informal support providers. The

Journal of Sex Research, 56(8), 1045-1057.

O'Driscoll, C., & Flanagan, E. (2016). Sexual problems and post-traumatic stress disorder

following sexual trauma: A meta-analytic review. Psychology and Psychotherapy: Theory,

Research and Practice, 89(3), 351-367.

V2 10/10/22

Weaver, T. L. (2009). Impact of rape on female sexuality: Review of selected literature. Clinical Obstetrics and Gynecology, 52(4), 702-711.

Zarski, A. C., Berking, M., Fackiner, C., Rosenau, C., & Ebert, D. D. (2017). Internet-based guided self-help for vaginal penetration difficulties: results of a randomized controlled pilot trial. The journal of sexual medicine, 14(2), 238-254.

V2 10/10/22